CLINICAL TRIAL: NCT05801406
Title: From Benchmark to Surgical Activity: the Role of Endobronchial Fiducial Markers for Ground Glass Lung Nodules Resection.
Acronym: Vortex_US
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, bandelli, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: IRCSS AOU Bologna
Record Dates: First submitted 2023-03-25; First posted 2023-04-06 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer; Lung Non-Small Cell Carcinoma; Lung; Node
Keywords: Ultrasound; Marker; Fluoroscopy; Lung; Cancer; Bronchoscopy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Tornado (Cook) — Fiducial marker endobronchial positioning under augmented fluoroscopy to mark ground glass opacities.

SUMMARY:
With the risen popularity of low-dose computed tomography (LDCT) for lung cancer screening, many patients present with peripheral pulmonary ground-glass nodules (GGNs) with a suspicious solid part. The appropriate diagnostic and management strategy for those lesions can be questionable. If malignancy is suspected, a surgical biopsy with the guidance of various localization methods available is recommended.

Each localization method has its advantages and disadvantages. Therefore, it may not be possible to establish a gold standard for localizing indeterminate lung nodules since comparative clinical trials are lacking.

DETAILED DESCRIPTION:
The management of pulmonary ground-glass nodules (GGNs) may be different. If GGN is an incidental finding through LDCT, the lesion should be followed according to the current guidelines. It is recommend a multidisciplinary team discussion to be initiated if a new solid component develops or the solid portion size grows on follow-up CT as the risk of malignancy is high. Attempts to preoperatively biopsy solid components in part-solid GGNs are often not feasible and not helpful in clinical settings. Currently, if malignancy is suspected, a surgical biopsy with the guidance of various localization methods is recommended. If malignancy is confirmed, sub-lobar resection may provide an excellent oncologic outcome.

The LungVision system is a novel augmented-fluoroscopy-based real-time navigation and guidance technology for bronchoscopy that can enable real-time visualization and localization of pulmonary nodules.

In this study, all patients over the age of 18 will be enrolled in case of finding of lung GGNs with the presence of a solid part inside> = 6 mm or with a solid part even less than 6 mm but with an increase in size. These must be subject to surgical treatment for both diagnostic or therapeutic purposes. These nodules must have a bronchus sign inside. In these patients, a bronchoscopy under general anesthesia with oro-tracheal intubation with LungVision system and r-EBUS will be performed to select the area to mark with fiducial marker. After fiducial marker placement, a CT scan will be performed to control the position of fiducial marker compared to the lesion. Patients will subsequently undergo surgical treatment by using intraoperative ultrasonography to detect the position of fiducial marker in the completely deflated lung. The correct positioning of the fiducial marker compared to the lesion and the complete surgical excision of the target lesion will be evaluated on the surgical specimen.

ELIGIBILITY:
Inclusion Criteria:

* all patients over the age of 18;
* lung GGNs with the presence of a solid part inside > = 6 mm or with a solid part even less than 6 mm but with an increase in size;
* subjects evaluated for surgical treatment during multidisciplinary tumor board.

Exclusion Criteria:

* Patients not eligible for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, all patients over the age of 18 will be selected in case of finding of lung GGNs with the presence of a solid part inside > = 6 mm or with a solid part even less than 6 mm but with an increase in size. These must be subject to surgical treatment for both diagnostic or therapeutic purposes.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events | 12 months
  Rate of complications due to endobronchial positioning of fiducial markers under augmented fluoroscopy to mark ground glass opacities.

SECONDARY OUTCOMES:
Number of fiducial markers completely removed | 12 months
  Number of fiducial markers placed under augmented fluoroscopy completely removed (margins free from disease) after surgical removal of ground glass opacities in the lung

CONTACTS AND LOCATIONS:
Overall Officials: Gian Piero Bandelli, MD, Principal Investigator — AOU Bologna - Italy
Locations (1):
- Gian Piero Bandelli, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Undecided